CLINICAL TRIAL: NCT06191497
Title: The Effect of Nicotine Exposure on Periodontal Tissues After Non- Surgical Periodontal Therapy With and Without the Use of a Chlorhexidine-based Antiseptic in Patients With Periodontitis
Brief Title: The Effect of Smoking and Chlorhexidine on Periodontal Tissues After Non- Surgical Periodontal Therapy in Patients With Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Aleksandar Pupovac, Assistant, Department of Periodontology, University of Rijeka
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHX 01/22
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Smoking; Periodontitis; Periodontal Diseases
MeSH Terms: conditions — Smoking; Periodontitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-smokers (Active Comparator): 15 non-smoking subjects with diagnosed periodontitis. All of them underwent NSPT
  Interventions: Procedure: non surgical periodontal therapy
- Non-smokers+ CHX (Experimental): 15 non-smoking subjects with diagnosed periodontitis. All of them underwent NSPT and used 0.12% chlorhexidine mouthwash for 15 days after therapy
  Interventions: Procedure: non surgical periodontal therapy; Drug: Chlorhexidine mouthwash
- Smokers (Active Comparator): 15 cigarette smoking subjects with diagnosed periodontitis. All of them underwent NSPT
  Interventions: Procedure: non surgical periodontal therapy
- Smokers + CHX (Experimental): 15 cigarette smoking subjects with diagnosed periodontitis. All of them underwent NSPT and used 0.12% chlorhexidine mouthwash for 15 days after therapy
  Interventions: Procedure: non surgical periodontal therapy; Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Procedure: non surgical periodontal therapy — NSPT based on Guided biofilm therapy principle (EMS Dental, Switzerland)
Drug: Chlorhexidine mouthwash — 0.12% chlorhexidine based mouthwash used twice a day for 15 days after therapy
  Arms: Non-smokers+ CHX; Smokers + CHX

SUMMARY:
The aim of this study is to evaluate whether the use of a chlorhexidine based oral antiseptic will improve clinical results of non-surgical periodontal therapy (NSPT) in smokers with periodontitis.

A randomized controlled clinical trial will be carried out on 60 subjects with periodontitis- 30 smokers and 30 non-smokers. All subjects will be clinically examined. The following periodontal indices will be measured: Full mouth plaque score (FMPS), Full mouth bleeding score (FMBS), Pocket probing depth (PPD), Clinical attachment level (CAL), Gingival recession (GR) and Tooth mobility (TM). All subjects will have NSPT carried out. Half of the subjects in each group will use a 0.12% chlorhexidine based mouth rinse twice a day during 15 days. Clinical examination will be repeated 8 weeks after NSPT and compared.

DETAILED DESCRIPTION:
A total of 60 subject will be recruited among patients seeking periodontal treatment at the Department. All subjects will have periodontitis diagnosed according to the criteria outlined in the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions. The subjects will be divided into two groups based on smoking status. The first group of 30 subjects will consist of cigarettes smokers and the second group of 30 non- smokers. All the subjects in the first group smoke for a minimum of 3 years and at least 10 cigarettes a day. Patients smoking e-cigarettes, tobacco heating systems, cigarettes without filter and occasional smokers will be excluded from the study. Moreover, minors, pregnant woman, patients with systemic diseases affecting periodontal tissues, immunodeficient patients, patients who used antibiotics in the previous six months, patients with orthodontic appliances or retainers and patients who previously had periodontal therapy or were in supportive therapy will be excluded from the study. A randomization plan based on sex (male; female), age (</> 50 years), nicotine exposure (smoker; non-smoker) and intervention (with/ without CHX) will be made using an online randomization software. All subjects will undergo a clinical examination before and 8 weeks after non-surgical periodontal therapy. Clinical examination will include all teeth except third molars and will be carried out using a millimeter graduated PCP-15 UNC periodontal probe (Hu-Friedy, Chicago, USA). The following periodontal indices will be measured: Full mouth plaque score (FMPS), Full mouth bleeding score (FMBS), Pocket probing depth (PPD), Clinical attachment level (CAL), Gingival recession (GR) and Tooth mobility (TM).

All subjects will have non-surgical periodontal therapy carried out according to the principles of Guided biofilm therapy (GBT) (EMS Dental, Geneve, Switzerland) using AIRFLOW Prophylaxis Master ultrasonic instruments (EMS Dental, Geneve, Switzerland) and Gracey curettes (Hu- Friedy, Chicago, USA). Moreover, half of the subjects in each group, 15 smokers and 15 non-smokers, will use a 0.12% chlorhexidine-digluconate based mouthwash (Curasept ADS 212, Curasept SpA, Saronno, Italy) twice a day for one minute during a period of 15 days. Subsequently, four subgroups of 15 subjects will be formed- non-smokers (NS), non-smokers who used CHX (NS-CHX), smokers (S) and smokers who used CHX (S-CHX).

ELIGIBILITY:
Inclusion Criteria:

* patients with periodontitis smokers and non smokers.

Exclusion Criteria:

* minors, pregnant woman, patients with systemic diseases affecting periodontal tissues, immunodeficient patients, patients who used antibiotics in the previous six months, patients with orthodontic appliances or retainers and patients who previously had periodontal therapy or were in supportive therapy
* Patients smoking e-cigarettes, tobacco heating systems, cigarettes without filter and occasional smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Full mouth plaque score | 8 weeks
  plaque accumulation
Full mouth bleeding score | 8 weeks
  gingival bleeding
Pocket depth | 8 weeks
  periodontal pocket depth in mm
Clinical attachment level | 8 weeks
  clinical attachment loss in mm
Gingival recession | 8 weeks
  gingival recession in mm
Tooth mobility | 8 weeks
  tooth mobility- Miller class

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dental medicine, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No
only data not affecting participants personal data will be shared upon reasonable request